CLINICAL TRIAL: NCT07372456
Title: The Effect of Nurse-Led Social Emotional Learning Program on Adolescents' Bullying, Victimization, and Bystander Behaviors
Brief Title: Nurse-Led Social Emotional Learning Program for Reducing Bullying, Victimization and Bystander Behaviors in Adolescents
Acronym: Nurse-Led SEL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Collaborators: Marmara University, Scientific Research Projects Committee (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 28.06.2024- 68
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Bullying Victimization; School Bullying; School Health; School Based Intervention
Keywords: Peer bullying; School health; Social emotional learning; Nurse; Middle school students; Nurse-Led intervention; Peer relationships; Adolescents

STUDY DESIGN:
Intervention Model Description: This study is parallel group randomized controlled study.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Students in the experimental group will participate in a structured six-week nurse-led social emotional learning intervention. The program comprises animations, an website, and a variety of learning activities designed to enhance emotional and social skills.
  Interventions: Other: Nurse-Led Social Emotional Learning-Based Education Program
- Control Group (No Intervention): Students in this group will continue their routine school curriculum without receiving the SEL-based program.

INTERVENTIONS:
Other: Nurse-Led Social Emotional Learning-Based Education Program — The Social Emotional Learning-Based Education Program will be implemented in the intervention group once a week for six weeks. The program was developed based on the principles of social emotional learning. Each week addresses one of the five core components of social emotional learning: self-awareness, self-management, responsible decision-making, relationship skills, and social awareness. The education will be delivered using various instructional methods, including lectures, problem-solving, question-and-answer, group discussions, case studies, scenario-based learning, gamification, and brainstorming. A range of audio-visual materials will be utilized, such as computers, projectors, presentation screens, speakers, remote controls, posters, brochures, videos, colored papers, educational booklets, and magazines. Additionally, scenarios prepared for the education program have been transformed into animations, and a dedicated website has been developed to support the intervention.
  Other Names: Nurse-Led SEL Program; NLSEL
  Arms: Intervention Group

SUMMARY:
This randomized controlled trial will evaluate the effect of a nurse-led social emotional learning (SEL) program on bullying, victimization, and bystander behaviors among adolescents. The study will be conducted in two public middle schools in Istanbul, Türkiye, with students in grades 6-8. Participants in the intervention group will receive structured SEL sessions designed to enhance emotional regulation, empathy, and problem-solving skills, while the control group will continue with routine education. Outcomes will be measured using validated scales at baseline, three months, and six months after the intervention.

DETAILED DESCRIPTION:
School violence is observed at all levels of education, but it is particularly prominent during middle school, which coincides with early adolescence. While violence tends to increase in primary school and decrease in higher grades of high school, no significant differences are observed between grade levels in middle school. Bullying has multiple negative consequences: for perpetrators, it is associated with suicide, weapon carrying, substance use disorders, and a tendency toward violence and criminal behavior in adulthood; for victims, it is linked to low self-esteem, anxiety disorders, and suicide. Due to these multifaceted negative effects, bullying prevention programs must be implemented as public health interventions. This study aims to evaluate the effect of a nurse-led, social emotional learning (SEL)-based education program on bullying, victimization, and bystander behaviors among adolescents attending grades 6, 7, and 8 in middle schools. Unlike many previous studies, this program not only seeks to reduce bullying and victimization but also aims to enhance bystander intervention. Furthermore, the intervention will be uniquely delivered by a nurse with a focus on fostering social emotional skills.This randomized controlled trial will be conducted between October 2025 and June 2026 in two public middle schools located in the Ümraniye district of Istanbul, Türkiye. The study will follow a pre-test, post-test, and follow-up test design with intervention and control groups. Randomization will be applied to ensure comparability, and participants with similar pre-test characteristics will be assigned to either group. The intervention group will receive the SEL-based training program, while the control group will continue with routine education. Post-tests will be conducted three months after the intervention, and follow-up assessments will be carried out at six months. Data will be collected in classrooms through face-to-face self-report surveys. Instruments include the Personal Information Form, Bullying Victimization Self-Efficacy Scale, Bullying and Cyberbullying Scale for Adolescents, Bystander Intervention in Bullying Scale, and Social Emotional Learning Skills Scale.Data entry will be performed electronically, and statistical analyses will be conducted using SPSS version 26. Tests appropriate for normal distribution will be used. A significance level of p < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in 6th, 7th, or 8th grade during the study period
* Students whose parents/legal guardians provide consent for participation
* Students who volunteer to participate in the study
* Students without communication barriers

Exclusion Criteria:

* Students who provide incomplete data in the pre-test, post-test, or follow-up assessments
* Students who do not fully participate in the intervention program
* Students with insufficient cognitive level to complete the study requirements

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-03-16 (Estimated); Study Completion 2026-06-08 (Estimated)

PRIMARY OUTCOMES:
Bullying and Cyberbullying Scale for Adolescents | Baseline (pre-test), 3 months (post-test), 6 months (follow-up)
  The Bullying and Cyberbullying Scale for Adolescents (BCS-A) was originally developed by Thomas et al. (2019) and adapted into Turkish by Özbey and Başdaş (2020). The scale consists of two parallel forms measuring bullying and victimization experiences of adolescents during the past three months. Each form includes four subscales: physical, verbal, relational, and cyber. The scale has 26 items in total. Subscale scores are calculated by dividing the sum of the items by the number of items in that subscale. Reported Cronbach's alpha values for the Turkish version range between 0.606-0.806 for the victimization subscale and 0.616-0.815 for the bullying subscale.
Bystander Intervention in Bullying Scale | Baseline (pre-test), 3 months (post-test), 6 months (follow-up)
  The scale was originally developed by Nickerson et al. (2014) to assess the level of bystander intervention in bullying situations. The Turkish adaptation was conducted by Demirbaş and Öztemel (2019). It consists of 16 items rated on a five-point Likert scale, covering five subdimensions: Noticing the Event, Interpreting the Event as Urgent, Accepting Responsibility to Help, Deciding How to Intervene, and Implementing the Decision to Intervene. Total scores range from 16 to 80, with higher scores indicating a greater likelihood of bystander intervention. Reported internal consistency (Cronbach's alpha) was 0.88 for the overall scale, 0.60 for Noticing the Event, 0.78 for Interpreting as Urgent, 0.67 for Accepting Responsibility, 0.75 for Deciding How to Intervene, and 0.78 for Implementing the Decision.

SECONDARY OUTCOMES:
Bullying Victimization Self-Efficacy Scale | Baseline (pre-test), 3 months (post-test), 6 months (follow-up)
  The Bullying Victimization Self-Efficacy Scale was originally developed by Kim et al. (2010) to assess students' self-efficacy in coping with bullying. The scale consists of 16 items across two subdimensions: Social Resources and Action. It is a five-point Likert-type scale (1 = Not sure, 5 = Very sure). The overall scale showed a Cronbach's alpha of 0.93. The Turkish adaptation was carried out by the researchers with a Cronbach's alpha of 0.88.
Social Emotional Learning Skills Scale | Baseline (pre-test), 3 months (post-test), 6 months (follow-up)
  The Social Emotional Learning Skills Scale was developed by Kabakçı and Owen (2010) based on the framework of social emotional learning. The scale consists of 40 items across four factors: Problem-Solving Skills, Communication Skills, Self-Enhancing Skills, and Coping with Stress Skills. It is a four-point Likert-type scale, with total scores ranging from 40 to 160. Higher scores indicate greater proficiency in social emotional learning skills. In the original reliability study conducted with 597 participants, Cronbach's alpha was 0.88 for the overall scale, 0.80 for Problem-Solving, 0.70 for Communication, 0.79 for Self-Enhancing, and 0.69 for Coping with Stress.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Ergun, Prof, RN, Study Chair — Marmara University; Esma Akgul, MSc, RN, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kabakçı, Ö. F., & Owen, F. K. (2010). Sosyal duygusal öğrenme becerileri ölçeği geliştirme çalışması. Eğitim ve Bilim, 35(157).
- [Result] Demirbaş, N. K., & Öztemel, K. (2019). Zorbalıkta seyirci müdahale ölçeği'nin (zsmö) Türkçe uyarlaması: geçerlik ve güvenirlik çalışması. Turkish Psychological Counseling and Guidance Journal, 9(54), 965-985.
- [Result] Nickerson AB, Aloe AM, Livingston JA, Feeley TH. Measurement of the bystander intervention model for bullying and sexual harassment. J Adolesc. 2014 Jun;37(4):391-400. doi: 10.1016/j.adolescence.2014.03.003. Epub 2014 Mar 24. PMID 24793386
- [Result] Ozbey H, Basdas O. Psychometric properties of the Turkish version of the Bullying and Cyber Bullying Scale for Adolescents (BCS-A). Psychiatry Res. 2020 Jul;289:112994. doi: 10.1016/j.psychres.2020.112994. Epub 2020 Apr 25. PMID 32408193
- [Result] Thomas HJ, Scott JG, Coates JM, Connor JP. Development and validation of the Bullying and Cyberbullying Scale for Adolescents: A multi-dimensional measurement model. Br J Educ Psychol. 2019 Mar;89(1):75-94. doi: 10.1111/bjep.12223. Epub 2018 May 3. PMID 29726005
- See also: Collaborative for Academic, Social, and Emotional Learning (CASEL). (2024a, May). Fundamentals of SEL — https://casel.org/fundamentals-of-sel/
- See also: Collaborative for Academic, Social, and Emotional Learning (CASEL). (2024b, May). What Is the CASEL Framework? — https://casel.org/fundamentals-of-sel/what-is-the-casel-framework/#social-awareness